CLINICAL TRIAL: NCT00056199
Title: Pilot Study of Intravitreal Injection of EYE001 (Anti-VEGF Pegylated Aptamer) for Advanced Ocular Disease of Von Hippel-Lindau (VHL) Disease
Brief Title: EYE001 to Treat Retinal Tumors in Patients With Von Hippel-Lindau Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030101; 03-EI-0101
Record Dates: First submitted 2003-03-07; First posted 2003-03-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Hippel-Lindau Disease
Keywords: Vision Loss; Optic Nerve Tumors; Macular Edema; Von Hippel-Lindau Disease; VEGF; EYE001; VHL
MeSH Terms: conditions — von Hippel-Lindau Disease; Vision Disorders; Optic Nerve Neoplasms; Macular Edema

INTERVENTIONS:
Drug: EYE001

SUMMARY:
This study will test the ability of the experimental drug EYE001 to reduce retinal thickening and improve vision in patients with Von Hippel-Lindau syndrome (VHL). Angiomas (blood vessel tumors) commonly develop in the back of the eye on the retina and the optic nerve in patients with VHL. Although the tumors are not cancerous, they may cause significant vision loss. Current treatments, including laser therapy, cryotherapy, and vitrectomy, may not be successful or possible for all patients. EYE001 decreases production of VEGF, a growth factor that is important for the formation of new blood vessels and that is elevated in VHL. Preliminary findings from studies of other retinal diseases suggest that EYE001 can reduce retinal thickening and improve vision.

Patients 18 years of age and older with retinal angiomas due to VHL in one or both eyes and central vision loss of 20/40 or worse may be eligible for this study. Participants will undergo the following tests and procedures:

* Medical history, physical examination, electrocardiogram (EKG) and blood tests.
* Eye examination, including eye pressure measurement and dilation of the pupils to examine the retina.
* Fluorescein angiography to evaluate the eye's blood vessels. For this test, a yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures will reveal if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Optical coherence tomography to measure retinal thickness. The eyes are examined through a machine that produces cross-sectional pictures of the retina. These measures are repeated during the study to determine changes, if any, in retinal thickening.
* Electroretinogram (ERG) to measure electrical responses generated from within the retina. For this test, the patient sits in a dark room for 30 minutes with his or her eyes patched. Then, a small silver disk electrode is taped to the forehead, the eye patches are removed, the surface of the eye is numbed with eye drops, and contact lenses are placed on the eyes. The patient looks inside an open white globe that emits a series of light flashes for about 20 minutes. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Stereoscopic color fundus photography to examine the back of the eye. The pupils are dilated with eye drops to examine and photograph the back of the eye.
* EYE001 injections to treat ocular angiomas. Patients receive EYE001 injections through a needle into the eye's vitreous (gel-like substance that fills the inside of the eye). Six injections are given over a 30-week period. Before each injection, the surface of the eye is numbed with anesthetic eye drops. This is followed by injection of another anesthetic into the lower portion of they eye in the clear tissue surrounding the white of the eye. After a few minutes, the EYE001 is injected into the vitreous. Patients receive EYE001 injections at the first visit (during enrollment) and again at 6, 12, 18, 24, and 30 weeks after the first injection.

At each injection visit, participants repeat most of the tests described above to evaluate the response to treatment and return a week later for another eye examination. After the last injection, patients whose vision has improved may receive three more treatments at visits 36, 42, and 48. All participants will return for examinations at week 54 and at 2 months after their final injection.

DETAILED DESCRIPTION:
Von Hippel-Lindau (VHL) is an autosomal dominant heritable disorder in which multiple benign and malignant neoplasms and cysts of specific histopathologies develop in the kidney, adrenal gland, pancreas, brain, spinal cord, eye, inner ear, epididymis, and broad ligament. Retinal angioma may be one of the earliest manifestations of VHL disease and may lead to a significant decrease in visual acuity of the affected individual. These tumors rarely regress spontaneously. The main cause of vision loss is retinal edema, specifically macular edema secondary to enlargement of peripheral retinal angiomas or angiomas found on or around the optic disk. Treatment of retinal angiomas depends on the location and size of the lesions but typically consists of photocoagulation or cryotherapy. However, there is no proven effective therapy for the treatment of VHL ocular lesions on or surrounding the optic nerve or lesions in the peripheral retina too large to respond to the traditional therapies. The genetic mutation found in VHL disease up-regulates the production of vascular endothelial growth factor (VEGF). Immunochemical studies of the VHL ocular lesions, as well as others found elsewhere in the body show marked increase in VEGF. This open-label study will pilot the use of anti-VEGF therapy (EYE001) in 5 patients to investigate the potential efficacy as a treatment for retinal angiomas associated with VHL. Patients will receive 6 intravitreal injections of study drug over a 30-week period, then return for a follow-up visit 1 year after initiating injections. The primary outcomes will be improvement in best corrected visual acuity of 15 letters or more at 1 year, reduction in retinal thickening and leakage at one year, changes in ERG amplitude and implicit time, and adverse events including local and systemic toxicities.

ELIGIBILITY:
INCLUSION CRITERIA:

Patient must understand and sign the informed consent.

Patient must be at least 18 years of age.

Patient must have retinal angiomas secondary to VHL in one or both eyes.

Patient must have either optic nerve tumors or peripheral tumors that have caused central vision loss of 20/40 or worse.

Patient must have clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography.

Patients must be post menopausal, surgically sterile for at least 12 months prior to study entry, or agree to use at least two effective forms of birth control.

All women of childbearing potential must have a negative serum pregnancy test at baseline and immediately prior to each injection and for at least 60 days following the last dose of EYE001.

Patient must have lab values indicative of adequate hematological function (hemoglobin greater than or equal to 10 g/dl, platelet count less than or equal to 130 x 10(9)/I, WBC 3.8-10.8 x 10(9)/I) within one month of baseline.

Patients must have lab values indicative of adequate liver function (serum bilirubin less than or equal to 1.5 mg/dl, SGOT/ALT, SGPT/AST, GGT and alkaline phosphotase within 2 x ULN) within one month of baseline.

Patients must have lab values indicative of adequate renal function serum creatinine less than or equal to 2.0 mg/dl and BUN within 2.0 x ULN within one month of baseline.

EXCLUSION CRITERIA:

Significant media opacities, including cataract that precludes quality fundus photographs of the posterior pole.

History or evidence of severe cardiac disease (electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within 6 months prior to baseline, atrial or ventricular tachyarrythmias requiring ongoing treatment).

History of stroke within 12 months of study entry.

History of or current acute ocular or periocular infection (including any history of ocular herpes zoster).

Any major surgical procedure within one month of study entry.

Known serious allergies to fluorescein dye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 2003-03; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Choyke PL, Glenn GM, Walther MM, Patronas NJ, Linehan WM, Zbar B. von Hippel-Lindau disease: genetic, clinical, and imaging features. Radiology. 1995 Mar;194(3):629-42. doi: 10.1148/radiology.194.3.7862955.
- [Background] Libutti SK, Choyke PL, Alexander HR, Glenn G, Bartlett DL, Zbar B, Lubensky I, McKee SA, Maher ER, Linehan WM, Walther MM. Clinical and genetic analysis of patients with pancreatic neuroendocrine tumors associated with von Hippel-Lindau disease. Surgery. 2000 Dec;128(6):1022-7;discussion 1027-8. doi: 10.1067/msy.2000.110239. PMID 11114638
- [Background] Manski TJ, Heffner DK, Glenn GM, Patronas NJ, Pikus AT, Katz D, Lebovics R, Sledjeski K, Choyke PL, Zbar B, Linehan WM, Oldfield EH. Endolymphatic sac tumors. A source of morbid hearing loss in von Hippel-Lindau disease. JAMA. 1997 May 14;277(18):1461-6. doi: 10.1001/jama.277.18.1461. PMID 9145719